CLINICAL TRIAL: NCT06133556
Title: Conditioning Regimen Containing Melphalan and Cladribine for Refractory / Relapsed AML
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIT2023023-EC-2
Record Dates: First submitted 2023-09-08; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control arm (Active Comparator): Busulfan/Cyclophosphamide, "standard" conditioning regimen as a control group. including Bu3.2mg/kg -5~-3d; Cy 80mg/kg，-2~-1d。 or alternative Bu/Cy regimen, Bu3.2mg/kg -9~-7d；Flu 30mg/m2 -6~-4d；Ara-C 2g/m2 -6~-4d；Cy 80mg/kg -3~-2d。
  Interventions: Drug: Bu/Cy regimen
- MCBC group (Experimental): using MCBC as conditioning regimen, Mel 60mg/ m2 -9~-8d, Cladribine 5 mg/m2 -9~-5d, Bu3.2mg/kg -5~-3d； Cy 30mg/kg -2~-1 d
  Interventions: Drug: MCBC regimen

INTERVENTIONS:
Drug: MCBC regimen — using MCBC as conditioning regimen, Mel 60mg/ m2 -9~-8d, Cladribine 5 mg/m2 -9~-5d, Bu3.2mg/kg -5~-3d； Cy 30mg/kg -2~-1 d
  Other Names: experiment group
  Arms: MCBC group
Drug: Bu/Cy regimen — control group, the standard conditioning regimen Busulfan/Cyclophosphamide
  Other Names: classic group
  Arms: control arm

SUMMARY:
This project is a prospective, multicenter, randomized controlled clinical study. The subjects were refractory / relapsed AML patients aged ≤ 60 years diagnosed by bone marrow cell morphology, immunology, genetics and therapeutic efficacy evaluation. The classical Bu / Cy scheme or MCBC scheme was used for pretreatment. The primary endpoint of the study was the 3-year recurrence-free survival rate after allogeneic hematopoietic stem cell transplantation, and the secondary endpoints were 3-year overall survival rate, recurrence rate, treatment-related mortality, and pretreatment-related toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Refractory / relapsed AML.
* Patients with a HLA matched related or unrelated donor (9~10/10) or haplo-identical related donor, plan to receive HSCT.
* Age ≤ 60 years old, men and women are not limited.
* The Eastern Oncology Collaborative Group Physical Status Assessment ( ECOG-PS ) was 0-2 points.
* Informed consent must be signed before the start of the study procedure. Informed consent must be signed by the patient or his or her immediate family members who are 18 years of age or older ; informed consent was signed by the legal guardian for children and adolescent patients under 18 years old. Considering the patient 's condition, if the patient 's signature is not conducive to the treatment of the disease, the informed consent is signed by the legal guardian or the patient 's immediate family.

Exclusion Criteria:

* Have a history of cancer and have received any treatment for this tumor in the past 3 years. But remove superficial bladder cancer, skin basal cells or squamous cell carcinoma, cervical epithelium. Intraepithelial neoplasia ( CIN ) or prostatic intraepithelial neoplasia ( PIN ).
* MPAL.
* It is known that the serological reaction of HIV or active hepatitis C virus is positive.
* The inability to cooperate with the requirements of research, treatment and monitoring due to mental illness or other conditions.
* Pregnant patients or patients who could not take appropriate contraceptive measures during treatment.
* Previously received hematopoietic stem cell transplantation.
* Active heart disease, defined as one or more of the following :

  1. ) Uncontrolled or symptomatic angina history.
  2. ) Myocardial infarction less than 6 months away from the study.
  3. ) Have a history of arrhythmia requiring drug treatment or severe clinical symptoms.
  4. ) Uncontrolled or symptomatic congestive heart failure ( > NYHA class 2 ).
  5. ) The ejection fraction is lower than the lower limit of the normal range.
* Researchers evaluated that is not suitable for the group.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 237 (Estimated)
Dates: Start 2023-11-24 (Estimated); Primary Completion 2028-10-20 (Estimated); Study Completion 2028-10-20 (Estimated)

PRIMARY OUTCOMES:
Relapse Free Survival | 3 year post-HSCT
  The AML relapse free survival post-HSCT

SECONDARY OUTCOMES:
Overall Survival | 3 year post-HSCT
  The overall survival post-HSCT
cumulative incidence relapse rate | 3 year post-HSCT
  cumulative incidence relapse rate post-HSCT
Non-relapse mortality | 3 year post-HSCT
  Non-relapse mortality post-HSCT
toxicity of conditioning regimen | 24w post-HSCT
  Adverse events as assessed by CTCAE to evaluate conditioning related toxicity
Immune reconstitution post-HSCT | 24w post-HSCT
  Using lymphocyte subset panel to assess immune recovery post-HSCT

IPD SHARING:
Plan to Share IPD: No